CLINICAL TRIAL: NCT07242521
Title: NON CANONICAL ACTIVATION OF BOOD COAGULATION (WORK PACKAGE 1) - VIE ALTERNATIVE DI ATTIVAZIONE DELLA CASCATA COAGULATIVA (PROGETTO 1)
Brief Title: NON CANONICAL ACTIVATION OF BOOD COAGULATION
Acronym: NCA-BC
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Prof. Giovanni Tinelli, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7843
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Oxidative Stress; vonWillebrand Disease; Carotid Artery Stenosis Symptomatic; Carotid Artery Stenosis Asymptomatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular diseases (CVD) are the major cause of mortality and morbidity worldwide and most of them are characterized by enhanced generation of active -thrombin (T) from the inactive Prothrombin zymogen (ProT), a reaction catalysed by factor Xa. CVD may be idiopathic, but also appear as the expression of thrombotic complications occurring with variable incidence and severity in different (apparently unrelated) diseases, such as for instance Type-2 Diabetes (T2D) , Chronic Kidney Disease (CKD), Inflammatory Bowel Disease (IBD) , Cancer , rheumatoid (RA) arthritis , autoimmune diseases such as the AntiPhospholipid Syndrome (APS), bacterial and viral infectious diseases, and amyloid-related diseases such as Alzheimer's disease, IgG light-chain amyloidosis and human transthyretin (hTTR) Senile Systemic Amyloidosis.This Project aims at combining different and complementary expertise with the general purpose of identifying new pathogenetic mechanisms for CVD and explored the possibility to devise novel and more effective therapeutic strategies.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the major cause of mortality and morbidity worldwide and most of them are characterized by enhanced generation of active -thrombin (T) from the inactive Prothrombin zymogen (ProT), a reaction catalysed by factor Xa. CVD may be idiopathic, but also appear as the expression of thrombotic complications occurring with variable incidence and severity in different (apparently unrelated) diseases, such as for instance Type-2 Diabetes (T2D) , Chronic Kidney Disease (CKD), Inflammatory Bowel Disease (IBD) , Cancer , rheumatoid (RA) arthritis , autoimmune diseases such as the AntiPhospholipid Syndrome (APS), bacterial and viral infectious diseases, and amyloid-related diseases such as Alzheimer's disease, IgG light-chain amyloidosis and human transthyretin (hTTR) Senile Systemic Amyloidosis. Globally, overall CVD affects >32% of people with T2D, being the major cause of mortality among T2D patients, with a mortality rate of about 50% [4]. Likewise, patients with IBD, a chronic and progressive inflammatory disease of the gastrointestinal tract, are increasing worldwide and have > 3-fold higher risk of venous thromboembolism (VTE) and portal venous system thrombosis, compared to general population, while necroscopy studies indicate that about 40% of patients that died with IBD had VTE [6]. Importantly, about 33% of patients with of severe bacterial sepsis by bothGram+ and Gram- are complicated by Disseminated Intravascular Coagulation (DIC), leading to multiple organ failure and death [10,11]. Very recently, the outbreak of the COVID19 pandemic has dramatically put forward the positive relation existing between thrombotic complications in SARS-Cov-2 infection and death [13]. Despite the receipt of anticoagulant thromboprophylaxis, in fact, critically ill patients with COVID19 present rates of VTE and arterial thrombosis of 15% and 30%, respectively, and autopsies revealed an incidence of deep venous thrombosis in 58% of non-survivors COVID19 patients. Importantly, the incidence of thrombogenesis is closely correlated with the high mortality observed in severe COVID19 cases, as 50% of non-survivors presented a pro-coagulant state, whereas only 7% of survivors were pro-coagulant [13]. Going from infectious to amyloid diseases, acquired SSA, an amyloidogenic pathology characterized by the deposition of hTTR deposits in the cardiac chambers of older patients, has been only recently recognized as a common, albeit underappreciated, cause of cardiomyopathy and heart failure in older adults, with an estimated total prevalence of 1-3% in elderly people >75 years of age.

For all these pathological settings, conventional thrombotic risk scores, such as the Framingham Risk Score [20], usually underestimate thrombotic risk [21] and, indeed, traditional risk factors for CVD (e.g., age, obesity, cigarette smoke, hypertension, dyslipidemia, hormonal therapy) have met limited success. Likely, this is caused by the intrinsically complex nature of the biochemical mechanisms leading to the generation of pathological clots, and the incomplete knowledge of the molecular links bridging, for instance, coagulation to other key physiopathological processes such as inflammation and innate immunity [11].

This Project aims at combining different and complementary expertise with the general purpose of identifying new pathogenetic mechanisms for CVD and explored the possibility to devise novel and more effective therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:Patients with carotid artery stenosis (CAS). One hundred patients with atheromatous carotid artery stenosis (CAS), admitted to the Unit of Vascular Surgery (RU-UniCATT) of Fondazione Policlinico Universitario A. Gemelli IRCCS for carotid endoarterectomy or stenting as per standard of care, will be enrolled. These patients will be divided into two cohorts composed of 50 patients each: 1) asymptomatic form of CAS (Cohort A) and 2) symptomatic CAS (Cohort B). In each cohort, T2DM and not diabetic patients will be enrolled with a 1:1 ratio. Patients on low-dose aspirin, statins, ACE inhibitors, metformin, pioglitazone, and sulfonylureas for DM patients.

Exclusion Criteria:any hemorrhagic coagulopathy, familial hypercholesterolemia, liver cirrhosis, sepsis, recent (12 months) surgery, trauma, IMA, or ischemic stroke, age <18 years old and inability to understand and sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid artery stenosis (CAS); asymptomatic form of CAS (Cohort A) and symptomatic CAS (Cohort B). In each cohort, T2DM and not diabetic patients will be enrolled with a 1:1 ratio.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Determination of total plasma protein carbonyls and VWF content and distribution of VWF multimers in T2D plasma samples. | six months
  Determination of total plasma protein carbonyls and VWF content and distribution of VWF multimers in T2D plasma samples. The total carbonyl content of plasma samples will be measured as stable markers of oxidative modification of proteins, using the ELISA Kit. VWF antigen (VWF:Ag), VWF as collagen binding activity (VWF:CBA), coagulation FVIII levels will be determined according to standard clinical assays.